CLINICAL TRIAL: NCT05259254
Title: Effectiveness, Feasibility, And Usability Of Mobile Application To Improve Adherence To Tuberculosis Treatment
Brief Title: Effectiveness Of Mobile Application To Improve Adherence To Tuberculosis Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mohd Fazeli bin Sazali (Other)
Collaborators: Ministry of Health, Malaysia (Other Government)
Responsible Party: Sponsor-Investigator, Mohd Fazeli bin Sazali, Principle Investigator, Universiti Malaysia Sabah
Organization: Universiti Malaysia Sabah (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PatuhTB01
Record Dates: First submitted 2022-02-17; First posted 2022-02-28 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Tuberculosis
Keywords: tuberculosis; adherence; mobile application
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Intervention Model Description: Following the diagnosis of TB by physician, patients will be directed to take daily medication of antiTB drugs. Patients will be randomised to two different groups of intervention which are standard directly observed therapy (DOT) and mobile application DOT.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Direct Observed Therapy (DOT) (Placebo Comparator): After a patient was diagnosed with TB, they will be provided TB therapy which is consist of health education and anti-TB medication. Patient that is not in life-threatening condition typically will be treated as outpatient. Patient will receive medication that will be monitored closely through DOT, which is either by health facilities (by healthcare staff), or community (by family members or community members). Observation of medication will be conducted daily, and the health care staff will sign the DOT diary provided to the patient to verify the medication consumption.
  Interventions: Other: Direct Observed Therapy
- Mobile application DOT (Active Comparator): The mobile application will be consisting of four basic modules which are: 1) reminder system, 2) visual observed therapy, 3) feedback, and 4) health education. Researcher will teach patient on how to record, and send video of every dose of medication ingested every day. Participants also required to show their mouth is empty by opening their mouth and sticking out their tongue. The participants also are required to record and send the self-recorded video of ingesting the medication daily. Researcher will subsequently view the video through a password protected website. The observation of taking medication will be completed until the end of study period.
  Interventions: Other: Mobile Application

INTERVENTIONS:
Other: Mobile Application — the mobile application will be consist of 4 modules which are: video observed therapy, health education, reminder system, and feedback.
  Arms: Mobile application DOT
Other: Direct Observed Therapy — it is a specific strategy that require identification, training, and supervision by various parties such as healthcare worker, community volunteer, or family members to directly monitor the ingestion of anti-TB medication. DOT was aimed to improve medication adherence by active monitoring and documenting the consumption of each dose taken. Conducting DOT is not only limited to directly observe the treatment, but also can assess medication side effects as well as to document the visit and information regarding medications (e.g., frequency and timing of taking medication).
  Arms: Standard Direct Observed Therapy (DOT)

SUMMARY:
Tuberculosis (TB) is a major public health concern, where it is among the top ten causes of death and the leading cause of death due to a single infectious agent globally. Providing standard anti-TB therapy for at least six months is recommended as one of the important strategies to control TB epidemic. However, prolonged duration of TB treatment raised issues of non-adherence. Non-adherence to TB therapy could negatively affect clinical and public health outcomes. Introduction of Direct Observed Therapy (DOT) has been used as a standard strategy to improve anti-TB adherence. Nonetheless, the DOT approach has been criticized due to inconvenience, stigma, reduced economic productivity, and reduced quality of life which ultimately could complicate the adherence issues. Apart from that, its effectiveness is debatable. Therefore, digital adherence technology could be an important alternative to DOT. Incorporation of Health Belief Model into the development of digital technology could potentially help to change behaviour and improve medication adherence. Hence, this study aimed to determine the effectiveness, feasibility, and usability of mobile application in improving TB medication adherence. This study proposed to conduct a pilot study to assess feasibility and usability followed by randomized, open-label, control trial among TB patients receiving TB care in several public health clinics in Kota Kinabalu, Putatan, and Penampang, Sabah, Malaysia. The eligible sample will be randomly assigned into mobile application DOT arm (intervention arm) and standard DOT arm (control arm). The primary outcome for this study is the successful completion of 80% or more of treatment observations that was scheduled in the two months following randomization. The secondary outcome measures are continuous variables including health related quality of life (HR-QOL), satisfaction level, and employment status. Multiple logistic regression analysis will be used to determine factors associated with primary outcome. Intention to treat and restricted analysis will be conducted. Independent sample t-test and repeated measures ANOVA will be used to compare the continuous secondary outcome between two intervention arms. The findings from this study are hopefully could provide insight into rethinking TB care delivery in order to achieve better TB treatment outcome.

DETAILED DESCRIPTION:
Background Tuberculosis (TB) is an infectious disease that is caused by a bacterium called Mycobacterium tuberculosis. Worldwide, TB is considered as one of the major public health threats, where it is among the top ten causes of death and a leading cause of death due to a single infectious agent. Even though the most form of TB infection are treatable, and death is preventable, World Health Organization (WHO) estimated that 10 million people were infected and fell ill due to TB infection in 2019 and causing death to 1.2 million people. In addition, TB infection was identified as the number one cause of death among people living with HIV, where it was estimated 208 000 deaths or approximately 40% among HIV positive individuals died due to TB infection.

TB infection and the death is preventable using a standard 6 months medication regime. However, long duration of anti-TB treatment posed significant challenges to TB patients. Non-adherence to anti-TB therapy is one of the major challenges in TB management. A recent study in South Africa estimated that treatment loss is mainly occurred at the point of treatment completion, with only 53% of overall TB cases are able to complete treatment. Failure to complete anti TB therapy can lead to poor treatment outcome, such as the increased risk of relapse, acquired drug resistant TB, treatment failure, progression of disease leading to complication, risk of death, and ongoing transmission of disease in the community.

Adherence to TB therapy is critical for the success of TB treatment. Adherence to TB therapy is multidimensional, which is comprised of five factors, namely socioeconomic factor, health system factor, condition-related factor, therapy-related factor, and patient-related factor.

Ending TB epidemic is one of the main target under the Sustainable Development Goals (SDG) which require a holistic approach that combines biomedical, public health, social, and economic intervention. Therefore, tackling the issues of non-adherence to TB therapy and follow-up requires a concerted effort from a wide range of social determinants of TB disease. Under the End TB strategy, it encompassed a comprehensive package of intervention, which consists of three pillars. The first pillar emphasized on the integrated, patient-centered care and prevention, which require the need to strengthen and expand the core functions of TB programs. It involves the need to embrace the new strategies and technologies to enhance patient care.

The expansion of mobile phone and internet access to various parts of the world has provide a good opportunity to incorporate the utilization of digital technology into public health practice. According to the global report by Global System for Mobile Communication Association (GSMA), almost half of world's population or 3.5 billion individuals are connected to the internet, where more than half of people in low middle-income country has been using mobile phone as the primary mean of internet access. Even though affordability, low level of digital literacy and skills, and perceived lack of relevance might serve as a barrier in the use of mobile phone, the gap in the usage of mobile phone has been decreased from 24% to 10% worldwide, which mainly contributed by increased affordability and internet access. Department of Statistics Malaysia (DOSM) reported that in 2019, 98% of Malaysian populations are using mobile phone. Among those who are using mobile phone, the smartphone users have been substantially increased from 89% in 2018 to 91% in 2019. High usage of mobile phone and internet connectivity among Malaysian population may provide an opportunity for an alternative strategy in enhancing the prevention and care of TB patients.

The utilization of digital technology to enhance adherence to TB therapy is particularly important and relevant to rethinking TB care delivery. In public health perspectives, enhancing adherence to anti-TB therapy can help to prevent relapse, drug resistance, and TB transmission in the community. A large nested case control study in Vietnam has found that one of the important predictors of TB recurrence is incomplete adherence to anti-TB therapy. In addition, TB care has been associated with negative consequences, especially in social and financial burden, not only because of the disease itself, but more importantly because of the treatment. Current strategy of Direct Observed Therapy (DOT) to ensure adherence of patients to TB treatment might cause problems to patients, as they are required to come to health facilities in daily manner to take the medication. Frequent visits to health clinic could cause disruption to their work, reduce productive time, and increase the risk of job insecurity. Furthermore, the disease is mostly affecting the age group with high economic productivity. Daily visits to healthcare facilities also could cause inconvenience to patients due to increase in travel time, waiting hours, and reduced participation in social activities . In addition, the disease and treatment itself also can cause a significant impact on a patient's life, such as quality of life, physical, psychological, and emotional wellbeing.

The use of digital technology in TB care provides an alternative in managing TB. When Direct Observed Therapy (DOT) has been introduced and implemented as one of the key strategies to improve adherence to TB therapy in the early 1990s, little consideration is taken to look at the needs of patients, especially among those who are economically productive. According to a recent systematic review, it was showed that DOT's effectiveness is varied compared to self-administered therapy. For example, DOT by family members was found to be not superior in improving treatment outcomes compared to self-administered therapy. However, institutional DOT provided for latent TB infection was found to be effective in improving treatment completion. The finding is consistent with another systematic review, which found that treatment success was low and intervention using DOT was not substantially improving treatment success. The use of digital technology in increasing adherence to TB therapy could help to reduce inconvenience to patients because of travelling to health facilities, risk of hospital acquired infection among visitors in health facilities and reduces the burden of supervision on healthcare workers.

Digital adherence technology might have several advantages over conventional strategy in TB care, especially using DOT. In a randomized clinical trial involving TB patients in UK, it has found that the use of video observed therapy (VOT) was an effective approach in TB therapy observation compared to DOT. VOT also was found to be the preferred method in treatment observation across a broad range of settings, providing a more acceptable, effective, and cheaper option for supervision of daily and multiple daily doses than DOT. In addition, VOT also a better option as it was proven in reducing observation time, reduced cost incurred because of observation, user's preference, and better psychosocial impact.

1.3 Justification Lack of adherence to anti-TB medication has been found to be associated with acquired drug resistance, TB relapse, TB complication, treatment failure, and ongoing transmission of disease in community. Implementation of digital adherence technology, such as using the mobile application can potentially improving medication adherence. However, many of these technology were lacking in incorporation of behavioral change model in their planning and development stage which explains the disappointing outcomes of many digital technology products. It is very important to understand that medication adherence is closely related to human behavior and motivation, and adoption of behavioral change theory into intervention can potentially affect medication adherence and ultimately improving treatment success. Thus, this study intended to adopt the Health Belief Model, one of the most common behavioral change theories into development of mobile application.

Digital adherence technology has been tested in various countries in the past and it was found to be varied in effectiveness, possible because of differences in settings, situation, user's belief, and knowledge. Thus, adopting the digital adherence technology in improving medication adherence would be tailored to Malaysian settings that is diverse in sociocultural background and beliefs. Studying the effectiveness of this technology in local population could provide knowledge to develop strategies to improve medication adherence and treatment success in the TB control program. Furthermore, there was no published study that was conducted among TB patients in Malaysian settings to identify the level of TB adherence as well as its effectiveness of various interventions in randomized clinical trials.

Research hypothesis:

1. There are no significant differences in proportion of participants receiving >80% of their total planned dose of medications in the 2 months following the randomization in between mobile application DOT with standard DOT users.
2. There are no significant differences in health-related quality of life mean score in between mobile application DOT with standard DOT group.
3. There are no significant differences in mean participants satisfaction score in between mobile application DOT with standard DOT group.
4. There are no significant differences in mean time loss due treatment observation between mobile application DOT and standard DOT group.
5. There are no significant differences in mean income loss due to treatment observation between mobile application DOT and standard DOT group.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed and all existing TB cases in maintenance phase.
* Age 18 years old and above
* Receiving standard therapy of daily antituberculosis drug according to Malaysian Clinical Practice Guideline of Tuberculosis 3rd Edition 2011.

Exclusion Criteria:

* No access to smart phone
* On injectable type of anti-TB
* Less than two months remaining in current treatment regime.
* Not planned to continue follow ups in study location in the next two months.
* Patients with psychiatric problem and no family members to assist taking medication at home.
* Not being able to understand Malay and English language
* Patients that health care staff consider needed intensive face-to-face support for emotional, medical, or structural reasons, as well as imminent risk of loss to follow up.
* Unconsented to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-05-28 (Estimated); Study Completion 2023-05-28 (Estimated)

PRIMARY OUTCOMES:
Adherence Level assessed by number of participants completed daily medication observation | 2 months
  This primary measure of outcome is to assess the level of adherence to anti-TB treatment. Decision to use 80% as cut off point is based on previous literature which concluded that adequate adherence was defined by the threshold of 76% to 80% of intended dose taken. According to the Malaysian national tuberculosis guideline, if the interruption of medication less than 20% during maintenance phase, the treatment might be stopped, provided that if the sputum AFB smear is negative. Thus, 80% cut off point is selected as a proxy measures to determine adherence to medication. 80% and more is considered as high adherence and less than 80% is considered as low adherence to medication.

SECONDARY OUTCOMES:
Retention and Completion Rate assessed by number of active users of mobile application and number of participants who can complete intervention from the date of randomization | 2 months
  Retention rate can be calculated by (number of active users of mobile application across period of observation / total number of users at day 0 of observation) x 100.
  AND
  Rate of completion of the intervention. Can be calculated by (i.e., number of participants who can complete the intervention from training to uploading the video of medication consumption / total number of users recruited at day 0) x 100.
Usability Score assessed by validated English and Malay version of Usability Scale Questionnaire for the Assessment of Mobile Apps | 2 months
  Usability will be assessed using a validated English and Malay version of Usability Scale Questionnaire for the Assessment of Mobile Apps by John Brooke (1986) (original questionnaire) & Muhammad Fadhil (Marzuki et al., 2018) (Malay version questionnaire). Usability questionnaire is consisting of 10 items questionnaire using 5-points Likert scale from 0 (strongly disagree) to 5 (strongly agree). The overall score will be calculated from the summation of all items scores multiply with 2.5. The overall score will be ranged from 0 to 100. According to previous study by original author and Malay version of usability score (Marzuki et al., 2018), usability score of 68 and above was recommended to indicate good usability of mobile application. The Cronbach Alpha of Malay version of questionnaire was 0.85.
Health-related quality of life (HR-QOL) assessed by English and Malay Version of EUROQOL EQ5D-3L Questionnaire | 2 months
  HR-QOL will be assessed using a standardised EUROQOL EQ5D-3L instrument. The questionnaire was validated and available in Malay and English language. The questionnaire is consisting of two pages; the EQ5D descriptive system and EQ5D visual analogue scale (EQ-VAS). The EQ5D descriptive system comprises five dimensions including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Meanwhile, each of the dimensions has three levels of severity, namely no problem, mild to moderate, and severe problem. The respondents will be asked to indicate their current health status by checking the box against the most appropriate answer for each of the five dimensions. The EQ-VAS assess the respondent's self-rated health in term of the vertical visual analogue scale, where there are two endpoints which are labelled as 'the best health you can imagine' and 'the worst health you can imagine'.
Patient satisfaction assessed by the English and Malay Version of Short-Form Patient Satisfaction Questionnaire (PSQ-18) | 2 months
  participants will be assessed using the Short-Form Patient Satisfaction Questionnaire (PSQ-18), which was originally developed by Marshall and Hays (Marshall & Hays, 1994). PSQ-18 consists of eighteen items with seven dimensions, which measures general satisfaction (Item 3 and 17), technical quality (Item 2, 4, 6, and 14), interpersonal manner (Item 10 and 11), communication (Item 1 and 13), financial aspect (Item 5 and 7), time spent with a healthcare provider (Item 12 and 15), and accessibility and convenience (Item 8,9,16, and 18). A five-points Likert scale will be used to score the eighteen items.
Employment assessed by asking the total monthly household income and total time needed for medication observation | 2 months
  participants will be asked in two questions regarding their employment
  * Loss of income as the result of treatment observation. The participants will be asked to estimate how much he loss in previous week in Ringgit Malaysia (RM)
  * Missed time from paid/unpaid work as the result of treatment observation. The participants will be asked to estimate how much time he loss in the previous week in minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Mohd Fazeli bin Sazali, MD, MPH, Principal Investigator — Universiti Malaysia Sabah
Locations (1):
- Mohd Fazeli bin Sazali, Kota Kinabalu, Sabah, Malaysia

IPD SHARING:
Plan to Share IPD: No